CLINICAL TRIAL: NCT04123444
Title: Efficacy and Safety of 72-hour Infusion of Prostacyclin (1 Nanogram(ng)/Kilo(kg)/Minute(Min)) in Patients With Septic Shock Induced Endotheliopathy - a Multicentre Randomized, Placebo-controlled, Blinded, Investigator-initiated Trial"
Brief Title: Infusion of Prostacyclin (Iloprost) vs Placebo for 72-hours in Patients With Septic Shock Suffering From Organ Failure
Acronym: COMBAT-SHINE
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Jakob Stensballe, MD, PhD (Other)
Collaborators: Innovation Fund Denmark (Individual); Independent Research Fund Denmark (Industry)
Responsible Party: Sponsor-Investigator, Jakob Stensballe, MD, PhD, Sponsor, Rigshospitalet, Denmark
Organization: Rigshospitalet, Denmark (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: COMBAT-SHINE; 2019-001131-31 (EudraCT Number)
Record Dates: First submitted 2019-10-09; First posted 2019-10-11 (Actual); Last update posted 2024-05-07 (Actual); Status verified 2024-05

CONDITIONS: Septic Shock
MeSH Terms: conditions — Shock, Septic | interventions — Iloprost; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: Randomization in 2 parallel arms Adaptive phase 2b/3 trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Patient, investigator, outcome assessor and care provider will be blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Iloprost (Experimental): Patients randomized to active treatment (n=190 patients) will receive continuous infusion of iloprost for 72 hours after inclusion or until discharge to ward or death, whichever comes first.
  Interventions: Drug: Iloprost
- Placebo (Placebo Comparator): Patients randomized to placebo treatment (n=190 patients) will receive continuous infusion of placebo for 72 hours after inclusion or until discharge to ward or death, whichever comes first.
  Interventions: Drug: Isotonic saline

INTERVENTIONS:
Drug: Iloprost — Continuously infusion for 72 hours. treatment dose 1 ng/kg/min
  Other Names: Iloprost infusion
  Arms: Iloprost
Drug: Isotonic saline — Continuously infusion for 72 hours.
  Other Names: Isotonic saline infusion
  Arms: Placebo

SUMMARY:
The purpose of this trial is to investigate the efficacy and safety of continuous intravenous administration of low dose iloprost versus placebo for 72-hours, in up to a total of 380 patients with septic shock suffering from organ failure.

The study hypothesis is that iloprost may be beneficial as an endothelial rescue treatment as it is anticipated to deactivate the endothelium and restore vascular integrity in septic shock patients suffering from organ failure caused by endothelial breakdown, ultimately improving survival.

DETAILED DESCRIPTION:
Patients with the most severe type of sepsis, those with septic shock have a mortality rate between 30% to 45% due to multiple organ failure. The poor outcome of shocked patients, and especially those with sepsis, may by related to microvascular endothelial dysfunction. Evidence support that iloprost infusion significantly improved endothelial function and integrity,

The main objective in this trial is to investigate whether continuous infusion of lov dose iloprost at a dose of 1 ng/kg/min for 72-hours is safe and significantly reduce organ failure score in the intensive care unit (ICU) compared to infusion of placebo in patients with septic shock induced endotheliopathy (SHINE).

Patients that are eligible for this trial will be temporarily incompetent due to acute severe illness relating to septic shock, therefore informed consent will be obtained from a scientific guardian. Next-of kin and subsequently the patient will co-sign as soon as possible hereafter. During the trial, patient will be give continuous infusion of low dose iloprost or placebo for 72 hours as well as additional blood samples will be obtained daily for the first 72 hours. Follow up on organ failure, mortality and quality of life will be performed on dag 28 and 90.

This trial is conducted in accordance with the Helsinki 2 Declaration and International Council for Harmonisation of Technical Requirements for Pharmaceuticals for Human Use, Guideline for Good Clinical Practice (ICH-GCP) and in compliance with the protocol. As part of the quality assurance on-site monitoring visit will be performed by the an independent GCP-unit including source data verification. Standard Operation Procedure (SOP) to address protocol specific procedures such as data collection and adverse event reporting are developed.

The number of patients participating is based on a power calculation using the data on mean daily SOFA score from a recent randomized, double blind, placebo controlled clinical trial in patients with septic shock: Levosimendan for the prevention of acute organ dysfunction in sepsis (LeoPARD). If the true effect of the intervention is a reduction in mean daily SOFA score of 20% (relative) and providing the trial with 90% power to detect this difference at a significance level of 0.05 will require a sample size of 380 patients.

A pre-planned, blinded interim analysis will be performed after 200 patients have been included in the trial and followed for 90 days.

ELIGIBILITY:
Inclusion Criteria:

All the following criteria must be fulfilled:

1. Adult intensive care patients (age ≥ 18 years)
2. Septic shock defined according to the Sepsis-3 criteria:

   * suspected or documented infection
   * persisting hypotension requiring vasopressors to maintain a mean arterial blood pressure of 65 mmHg or above
   * Lactate level of 2 mmol/L or above despite fluid therapy within the last 3 hours at screening
3. Soluble thrombomodulin (sTM) above 10 ng/mL

Exclusion Criteria:

Patients who fulfil any of the following criteria will be excluded:

1. Withdrawal from active therapy
2. Pregnancy
3. Known hypersensitivity to iloprost.
4. Life-threatening bleeding as defined by the treating physician
5. Known severe heart failure (New York Heart Association (NYHA) class IV)
6. Suspected acute coronary syndrome
7. Previously included in this trial
8. Septic shock for more than 12 hours at the time of screening
9. Informed consent cannot be obtained
10. Included in other clinical trials with prostacyclin within 90 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 279 (Actual)
Dates: Start 2019-10-30 (Actual); Primary Completion 2022-06-28 (Actual); Study Completion 2022-06-28 (Actual)

PRIMARY OUTCOMES:
Modified Sequential Organ Failure Assessment (SOFA) | Up to 90 days after randomization
  Mean daily modified SOFA score in the intensive care unit (scores for each of five systems range from 0 to 4, with higher scores indicating more severe dysfunction; range score 0-20).

SECONDARY OUTCOMES:
28 and 90-day mortality | Day 28 and 90 after randomization
  Vital status of the patient at day 28 and day 90
Vasopressor free days | Until ICU discharge, maximun 90 days after randomization
  Days alive and without vasopressor at day 90.
Mechanical ventilation free days | Until ICU discharge, maximun 90 days after randomization
  Days alive and without invasive mechanical ventilation at day 90
Renal replacement free days | Until ICU discharge, maximun 90 days after randomization
  Days alive and without renal replacement therapy at day 90
Serious adverse reactions (SARs) | Until day 7 after randomization
  Numbers of patients with one or more serious adverse reactions (SARs) and total number of SARs
Serious adverse events (SAEs) | Until day 7 after randomization
  Numbers of patients with one or more and total number of serious adverse events and total number of SAEs; SAEs defined as ischaemic events and bleeding events (requiring more than 2 red blood cells (RBCs) within 24 hours or ongoing bleeding.

CONTACTS AND LOCATIONS:
Overall Officials: Morten Bestle, MD, PhD, Principal Investigator — Nordsjaelands Hospital
Locations (6):
- Denmark (6):
  - Dept. of Anaesthesia and Intensive Care, Bispebjerg Hospital, Copenhagen
  - Dept. of Intensive Care, Copenhagen University Hospital, Rigshospitalet, Copenhagen
  - Dept. of Intensive Care, Copenhagen University Hospital Herlev, Herlev
  - Dept. of Anaesthesia and Intensive Care, Nordsjaelands Hospital, Hillerød
  - Dept. of Anaesthesia and Intensive Care, Hvidovre Hospital, Hvidovre
  - Region Sealand University Hospital, Køge

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bestle MH, Stensballe J, Lange T, Clausen NE, Soe-Jensen P, Pedersen KH, Gybel-Brask M, Kjaer MN, Steensen CO, Jensen DB, Gartner R, Schonemann-Lund M, Kristiansen KT, Lindhardt A, Johansson PI, Perner A. Iloprost and Organ Dysfunction in Adults With Septic Shock and Endotheliopathy: A Randomized Clinical Trial. JAMA Netw Open. 2024 Sep 3;7(9):e2432444. doi: 10.1001/jamanetworkopen.2024.32444. PMID 39259541
- [Derived] Bestle MH, Clausen NE, Soe-Jensen P, Kristiansen KT, Lange T, Johansson PI, Stensballe J, Perner A. Efficacy and safety of iloprost in patients with septic shock-induced endotheliopathy-Protocol for the multicenter randomized, placebo-controlled, blinded, investigator-initiated trial. Acta Anaesthesiol Scand. 2020 May;64(5):705-711. doi: 10.1111/aas.13546. Epub 2020 Feb 3. PMID 31950481